CLINICAL TRIAL: NCT01747707
Title: Phase II Clinical Trial of Cisplatin,Docetaxel and S-1 as First Line Chemotherapy for Advanced Gastric and Gastroesophageal Junction Cancer
Brief Title: Cisplatin,Docetaxel and S-1 for Advanced Gastric and Gastroesophageal Junction Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Associate professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-31
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: gastric cancer; gastroesophageal junction cancer; chemotherapy; docetaxel; cisplatin; S-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Cisplatin; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel, cisplatin and S-1 (DCS) (Experimental): All patients receive the combination therapy of docetaxel, cisplatin and S-1 for a maximum of 6 cycles. Docetaxel 60mg/m2 IV infusion over 1 hour on d1; Cisplatin 30mg/m2 IV infusion on d1,2; S-1 40mg orally twice a day for patients with the body surface area (BSA) less than 1.25m2, 50mg twice a day with the BSA between 1.25 and 1.5m2, 60mg twice a day with the BSA over 1.5m2.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: S-1

INTERVENTIONS:
Drug: Docetaxel
  Other Names: taxotere
Drug: Cisplatin
Drug: S-1
  Other Names: TS-1

SUMMARY:
The combination of Cisplatin and S-1 (CS) achieved a response rate of approximately 45% with the PFS being around 6 months and overall survival time being 13 months in Japanese and Chinese gastric patients. It remains unclear whether the addition of docetaxel to CS would further enhance the efficacy as it dose in DCF(docetaxel, cisplatin and 5-fluorouracil). This is a single center, phase II clinical trial to evaluate the efficacy of docetaxel, cisplatin and S-1 (DCS) as first line chemotherapy for patients with advanced gastric and gastroesophageal junction cancer.

DETAILED DESCRIPTION:
This is a single arm trial. All Patients will receive up to 6 cycles of triple chemotherapy with docetaxel, cisplatin and S-1. Given the severe toxicity of DCF regimen, here the total dose of docetaxel and cisplatin is both reduced to 60mg/m2. For patients with CR/PR/SD disease after 6 cycles of chemotherapy, maintenance therapy with S-1 are recommended. Antitumor activity will be evaluated every two cycles according to RECIST1.1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable advanced gastric or gastroesophageal junction cancer;
* No previous chemotherapy and radiation for advanced disease except palliative radiation for a local pain control;
* At least one evaluable lesion per RECIST (Response Evaluation Criteria in Solid Tumors) 1.1;
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1;
* Recovery from the toxicities of previous therapy;
* Adequate bone marrow and organ function. Hb≥8 G/L; Absolute neutrophil ≥ 2.0 G/L; PLT ≥100 G/L ;ALT/AST ≤1.5 ULN or ≤5ULN with liver metastases; TBIL ≤1.5 ULN; Cr≤1.0 ULN;
* Life expectancy ≥3 months;
* For men and women of childbearing potential, agree on taking effective contraceptive method of birth control from the signed informed consent until 3 months after the last study drug administration;
* Signed informed consent.

Exclusion Criteria:

* Pathology type other than adenocarcinoma,such as squamous cell carcinoma;
* Previous treatment with taxanes, cisplatin or S-1;
* Relapse within 6 months after the end of adjuvant chemotherapy;
* Known brain metastases;
* Complete or incomplete intestinal obstruction or uncontrolled gastrointestinal bleeding;
* Known deficiency of DPD enzyme;
* Kown HIV infecton or drug addiction;
* Any acute or chronic medical or psychiatric condition that would make the patient inappropriate for entry into this trial in the judgement of investigators;
* Myocardial infarction within 6 months prior to the entry of this trial;
* Known history of allergic reaction to taxanes and platinum;
* Pregnant or breast feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
overall survival time (OS) | 14 months
  To determine the OS of DCS in patients with chemo-naive, advanced gastric or gastroesophageal junction cancer.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months
  To determine the PFS of DCS in patients with chemo-naive, gastric or gastroesophageal junction cancer
safety profile | 4 months
  To determine the tolerability of DCS in patients with chemo-naive, gastric or gastroesophageal junction cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, M.D, Principal Investigator — Cancer Hospital & Institute, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital & Institute, Chinese Academy of Medical Sciences, Beijing, China